CLINICAL TRIAL: NCT01584427
Title: ButCoIns - Metabolic Effects of Resistent Starch and Arabinoxylans in Subjects With Metabolic Syndrome
Acronym: ButCoIns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, AnneMarie Kruse, Professor Kjeld Hermansen, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CERN-ButCoIns
Record Dates: First submitted 2012-04-20; First posted 2012-04-25 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Metabolic Syndrome
Keywords: Dietary fibers; Resistent Starch; Arabinoxylans; Postprandial lipaemia; Insulin sensitivity; Body composition; Gene expression; Metabolic rate; Blood pressure
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Carbohydrate Diet (Active Comparator): 4 weeks of intervention with a diet rich in Arabinoxylans and Resistent Starch.
  Interventions: Dietary Supplement: Healthy Carbohydrate Diet vs. Western Style Diet
- Western Style Diet (Placebo Comparator): 4 weeks of intervention with a diet with low content of Resistent Starch and Arabinoxylans
  Interventions: Dietary Supplement: Healthy Carbohydrate Diet vs. Western Style Diet

INTERVENTIONS:
Dietary Supplement: Healthy Carbohydrate Diet vs. Western Style Diet — Cross over study with two intervention diets. Healthy Carbohydrate Diet with approximally 55 g of dietary fibers (arabinoxylan and resistant starch)compared with western style diet with low content of dietary fibers.

SUMMARY:
Background Life style related disease is an increasing problem all over the world. The Metabolic Syndrome (MetS) is a condition characterized by abdominal obesity, high blood lipids, high blood pressure and slightly elevated blood sugar. Subjects with MetS have high risk of developing Type 2 Diabetes and cardiovascular disease.

Dietary fibers have been shown to have positive effects on the components of MetS. The investigators have special interest in the combination of two types of fiber (Resistant (RS) starch and Arabinoxylans (AX)) .

Hypotheses Increase of RS and AX in the dietary composition has a positive effects on components of MetS i.e. decreases blood lipids, improves blood sugar, blood pressure and markers of inflammation.

The subjects undergo two dietary interventions of 4 weeks duration each: A "Healthy Carbohydrate Diet" with a high content of RS and AX is compared to a "Western Style Diet" with a low content of RS and AX.

DETAILED DESCRIPTION:
Background Life style related disease is an increasing problem all over the world. The Metabolic Syndrome (MetS) is a condition characterized by abdominal obesity, dyslipidemia, hypertension and impaired glucose tolerance. Subjects with MetS have high risk of developing Type 2 Diabetes and CVD.

Resistant Starch (RS) and Arabinoxylans (AX) are dietary fibers that have been shown to have positive effects on the components of MetS. The combination of RS and AX has not been tested before .

Hypotheses Increase of RS and AX in the dietary composition has a positive effects on components of MetS i.e. decreases postprandial lipaemia, improves glucose tolerance, insulin resistance, blood pressure and markers of inflammation.

Design:

A nonblinded randomized cross over study Two dietary interventions of 4 weeks duration each. A healthy carbohydrate Diet with a high content of RS and AX is compared to a Western Style diet with a low content of RS and AX. Between the two interventions, there is a wash out period of 4 weeks.

The primary outcome is postprandial lipaemia estimated by a high fat meal test of 6 hours duration. The test is performed before and after each intervention.

Secondary outcomes are:

* Glucose tolerance and insulin resistance estimated by OGTT
* 24 hours blood pressure
* MRI estimation of liver fat content
* Postprandial changes in genes of adipose tissue

ELIGIBILITY:
Inclusion Criteria: At least 3 out of the 5 following criterions

* Central obesity (Female >80 cm, Male >94)
* HDL cholesterol (female < 1,03 mmol/l, male < 1,29 mmol/l)
* Blood Pressure (> 130/85)
* Fasting Blood Glucose > 5,6 mmol/L

Exclusion Criteria:

* Diabetes
* Gastrointestinal disease
* Anticoagulation treatment
* Serious liver, heart or kidney disease
* Anaemia
* Corticosteroid treatment
* Waist circumference above 130 cm
* Alcohol or drug addiction
* Pregnancy og lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Postprandial triglycerides | 4 weeks
  Plasma Triglycerides are estimated during a high fat meal test of 6 hours duration. The test is performed before and after each intervention of 4 weeks.

SECONDARY OUTCOMES:
Change in insulin sensitivity | 4 weeks
  -Estimated by an OGTT where glucose and insulin are measured several times and insulin sensitivity is estimated according to the Matsuda Index. The test is performed before and after each intervention of 4 weeks.
Metabolic Rate | 4 weeks
  The metabolic rate is measured by indirect calometri (Deltatrac II) in the fasting state and two hours after ingestion of a fatty mixed meal. The test is performed before and after each intervention period.
Body composition | 4 weeks
  H-MRS of liver before and after intervention in order to estimate the fat content.
Twenty-Four-Hour Blood Pressure | 4 weeks
  Performed in the free-living situation. Data analysis are grouped in mean day, mean night and mean 24 h. Measured at baseline and at the end of each intervention.
Gene expression in adipose tissue | Four weeks
  Fat biopsies are take from abdominal adipose tissue and analyzed by real time PCR to see if gene expression changes after a high intake of dietary fiber.
Inflammatory Markers after 4 weeks of intervention | 4 weeks
  hs CRP, IL-6 and adiponectin are measured at baseline and at the end of each intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark